CLINICAL TRIAL: NCT02457962
Title: Mayo Clinic Radiotherapy Patient Outcomes Registry and Biobanking Study
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 15-000136
Record Dates: First submitted 2015-05-11; First posted 2015-05-29 (Estimated); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumors; Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Years
Biospecimen Retention: Samples With DNA — Blood specimens stored for use in future research with permission of participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To collect and analyze specimens that will correlate with clinical outcomes such as acute and late toxicities, quality of life, local control, and survival of patients treated with photon/proton therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Treated with photon/proton at Mayo Clinic Rochester in Radiation Oncology
2. Radiation therapy for curative intent

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients being treated at Mayo Clinic with photon/ proton therapy.
Sampling Method: Non-Probability Sample
Enrollment: 14266 (Actual)
Dates: Start 2015-04-23 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
analyze acute and late toxicities using CTCAE 4.03 | Patients will be followed for the duration of their life, an expected average of 20 years
analyze quality of life using LASA-3 and FACT-E | Patients will be followed for the duration of their life, an expected average of 20 years

SECONDARY OUTCOMES:
analyze local control through tumor assessments | Patients will be followed for the duration of their life, an expected average of 20 years
analyze survival by contacting patient and EMR (electronic medical record) review | Patients will be followed for the duration of their life, an expected average of 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Nadia N. Laack, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials